CLINICAL TRIAL: NCT01280110
Title: The Effects of BAK on the Blood Aqueous Barrier of Pseudophakic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Vital Paulino Costa, Professor of Ophthalmology, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VPC1
Record Dates: First submitted 2011-01-18; First posted 2011-01-20 (Estimated); Results first posted 2012-07-12 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Dry Eye Syndromes
Keywords: dry eye; pseudophakia; cornea; lubricating drop; BAK; blood aqueous barrier; blood-retina barrier
MeSH Terms: conditions — Dry Eye Syndromes; Pseudophakia; Corneal Diseases | interventions — Hypromellose Derivatives; Carboxymethylcellulose Sodium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preserved (BAK 0.006%) lubricating drop (Active Comparator): One group will receive preserved lubricating drops 4 times a day for 1 month.
  Interventions: Drug: Hydroxypropylmethylcellulose
- Preservative-free lubricating drops (Active Comparator): The second group will receive preservative-free lubricating drops 4 times a day for 1 month.
  Interventions: Drug: Carboxymethylcellulose

INTERVENTIONS:
Drug: Hydroxypropylmethylcellulose — 22 patients will receive this lubricating drop 4 times a day for 1 month
  Other Names: Retin Active
  Arms: Preserved (BAK 0.006%) lubricating drop
Drug: Carboxymethylcellulose — 22 patients will receive this lubricating drop 4 times a day for 1 month.
  Other Names: Optive UD
  Arms: Preservative-free lubricating drops

SUMMARY:
BAK is one of the most frequent preservatives in eye drops. BAK is a quaternary ammonium salt with surfactant qualities. It can be bacteriostatic or bactericidal depending on the concentrations used. It has been shown to be effective against most bacteria with a few exceptions, such as Pseudomonas aeruginosa, or picornaviruses. It as been widely used in eyedrops, nose sprays, hand and face washes, mouthwashes, spermicidal creams, and in various other cleaners, sanitizers, and disinfectants. BAK gained popularity when it was first introduced because it also enhances corneal penetration of some drugs by causing epithelial separation.

It is present in several ophthalmic formulations, including most of the antiglaucoma medications. If used chronically, BAK has been found to cause ocular surface changes, such as dry eye and punctuate keratitis. BAK has also been suggested to promote a break in the blood aqueous barrier, which may lead to undesirable consequences, such as uveitis and cystoid macular edema. However, this information is controversial. The purpose of this study is to evaluate the consequences of BAK on the blood-retinal and blood-aqueous barriers of pseudophakic patients receiving BAK-preserved lubricating drops.

DETAILED DESCRIPTION:
The primary hypothesis behind the study is that BAK may lead to a break in the blood-retina barrier in pseudophakic eyes, leading to an increase in macular thickness, compared to a non-BAK containing solution. The secondary hypothesis is that solutions containing BAK will increase the permeability of the blood aqueous barrier compared to non-BAK solutions. If the hypotheses are confirmed, they may serve as a contraindication to the use of BAK-preserved drops in pseudophakic eyes requiring chronic use of medications.

This is a prospective, randomized, examiner-masked, controlled study involving 44 pseudophakic eyes of 44 patients. Patients receiving any other eyedrop, with a previous history of uveitis, posterior capsule rupture or any other ophthalmic surgery will be excluded. Patients will be randomized to the use of a BAK-preserved lubricating drop or to the use of a non-preserved lubricating drop q.i.d for one month. Effects on the blood aqueous barrier will be objectively measured with a laser flare meter (Kowa, Japan) at baseline, 15 days and one month after inclusion. Patients will also have OCT images (Cirrus, Zeiss, USA) of the macula at the same time intervals to evaluate the possible effects on the blood-retina barrier. Macular thickness and the presence of cystoid macular edema will be evaluated at each time interval.

ELIGIBILITY:
Inclusion Criteria:

* Pseudophakic eyes that underwent cataract surgery at least 6 months before.

Exclusion Criteria:

* Use of any eyedrop.
* Other conditions associated with a break in the blood-aqueous or blood retina barrier (ie diabetes, ARMD, vasculitis, uveitis)
* Previous history of cystoid macular edema.
* Previous ocular surgery other than cataract surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vital P Costa, MD, Principal Investigator — Department of Ophthalmology, University of Campinas
Locations (1):
- Department of Ophthalmology, University of Campinas, Campinas, São Paulo, Brazil

REFERENCES:
- [Background] Baudouin C, Labbe A, Liang H, Pauly A, Brignole-Baudouin F. Preservatives in eyedrops: the good, the bad and the ugly. Prog Retin Eye Res. 2010 Jul;29(4):312-34. doi: 10.1016/j.preteyeres.2010.03.001. Epub 2010 Mar 17. PMID 20302969
- [Background] Noecker RJ, Herrygers LA, Anwaruddin R. Corneal and conjunctival changes caused by commonly used glaucoma medications. Cornea. 2004 Jul;23(5):490-6. doi: 10.1097/01.ico.0000116526.57227.82. PMID 15220734
- [Background] Ammar DA, Noecker RJ, Kahook MY. Effects of benzalkonium chloride-preserved, polyquad-preserved, and sofZia-preserved topical glaucoma medications on human ocular epithelial cells. Adv Ther. 2010 Nov;27(11):837-45. doi: 10.1007/s12325-010-0070-1. Epub 2010 Oct 7. PMID 20931366

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period started on March 2011 through December 2011 in the Department of Ophthalmology at the Hospital das Clínicas - State University of Campinas.
Period: Overall Study
Arm/Group | Preserved (BAK 0.006%) Lubricating Drop | Preservative-free Lubricating Drops
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preserved (BAK 0.006%) Lubricating Drop | Preservative-free Lubricating Drops | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 16 | 15 | 31
Age Continuous [Mean (Standard Deviation); unit: years] | 69 (10.7) | 65.2 (12.2) | 67.1 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 13 | 9 | 22
Region of Enrollment [Number; unit: participants]
  Brazil | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Aqueous Humor Flare
Description: Aqueous humor flare indicates the degree of a break in the blood-aqueous barrier. It is objectively measured with a Laser flare meter.
Time Frame: Baseline, 15 days and 30 days.
Population: Statiscal power of 80%.
Measure: Mean (Standard Deviation); unit: photons/msec
Groups:
- Preserved (BAK 0.006%) Lubricating Drop: One group will receive preserved lubricating drops 4 times a day for 1 month. The flare will be evaluated with Laser Flare Cell Meter (Kowa, FM 500, Japan). The patients will have 3 evaluations (baseline, 15 days and 30 days). The baseline measure is done before the use of the eyedrops.
- Preservative-free Lubricating Drops: he second group will receive preservative-free lubricating drops 4 times a day for 1 month. The flare will be evaluated with Laser Flare Cell Meter (Kowa, FM 500, Japan). The patients will have 3 evaluations (baseline, 15 days and 30 days). The baseline measure is done before the use of the eyedrops.
Arm/Group | Preserved (BAK 0.006%) Lubricating Drop | Preservative-free Lubricating Drops
Number analyzed (Participants) | 22 | 22
photons/msec
  Baseline | 8.4 (2.7) | 9.3 (2.6)
  15 days | 11.4 (5.1) | 8.4 (2.8)
  30 days | 11.9 (5.9) | 8.4 (2.5)

2. Secondary Outcome: Macular Thickness
Description: Macular thickness will be measured with an Optical coherence tomography (OCT). Measures 5% under the normal population according to the OCT software will be considered break in the blood-retina barrier.
Time Frame: Baseline, 15 days and 30 days.
Population: Statiscal power of 80%
Measure: Mean (Standard Deviation); unit: μm
Groups:
- Preserved (BAK 0.006%) Lubricating Drop: One group will receive preserved lubricating drops 4 times a day for 1 month. The central macular thickness was obtained through Cirrus™ HD-OCT (Zeiss). Mode 512x128 macular cube scan
- Preservative-free Lubricating Drops: The second group will receive preservative-free lubricating drops 4 times a day for 1 month. The central macular thickness was obtained through Cirrus™ HD-OCT (Zeiss). Mode 512x128 macular cube scan
Arm/Group | Preserved (BAK 0.006%) Lubricating Drop | Preservative-free Lubricating Drops
Number analyzed (Participants) | 22 | 22
μm
  Baseline | 258.5 (26.7) | 259.2 (26.8)
  15 days | 254.9 (24.2) | 256.4 (27.6)
  30 days | 255.9 (25.1) | 258.3 (29.1)

ADVERSE EVENTS:
Arm/Group | Preserved (BAK 0.006%) Lubricating Drop | Preservative-free Lubricating Drops
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No